CLINICAL TRIAL: NCT05777733
Title: The Effect of N_acetylcystein as an Antioxidant on Iron Overload and Frequency of Blood Transfusion in β-thalassemia Major Patients at Assiut Childern Hospital University
Brief Title: NAC Effect on Iron Overload and Blood Transfusion in β-thalassemia Major
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Adel Saber morsi, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: NAC as antioxidant
Record Dates: First submitted 2023-01-07; First posted 2023-03-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-03

CONDITIONS: Thalassemia Major
Keywords: N_acetylcystein antioxidant effect
MeSH Terms: conditions — beta-Thalassemia | interventions — N-monoacetylcystine

STUDY DESIGN:
Intervention Model Description: N-acetylcystein in dose 10mg /kg single oral dose will be given for 6 months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N_acetylcystein as antioxidant on iron and frequency of blood transfusion in thalassemia major (Experimental): N_acetylcystein administration on single oral dose 10mg /kg for 6 months and it's effect on iron and frequency of blood transfusion before and after its use.
  Interventions: Drug: n-acetylcystine

INTERVENTIONS:
Drug: n-acetylcystine — Single daily oral administration of N_acetylcystein on dose 10mg /kg/day
  Other Names: acetylcystein

SUMMARY:
The effect of N_acetylcystein as an antioxidant on iron overload and frequency of blood transfusion in β-thalassemia major patients at Assiut Childern Hospital University And its cosubmitted for partial fulfillment of master degree in Pediatrics

DETAILED DESCRIPTION:
Beta thalassemia major it menifests after 6 months of life by severe anemia requiring life-long blood transfusion,which is the the gold standard therapy causing many complications including iron overload which associated to a certain extent with the generation of labile iron in the pathological red blood cell (RBC). The appearance of such forms of iron at the inner and outer cell surfaces exposes the cell to formation of reactive oxygen species (ROS),particularly the hydroxyl radical (·OH) serving as a Fenton reagent, Hydroxyl radical facilitated by membraneassociated iron might be particularly harmful because radical generation would be relatively sequestered from the cell antioxidant capacity and occur directly adjacent to lipid and protein membrane components exceeding cellular defense capacities causing oxidtive stress with prematre cell damage which is the main pathophysiological process in thalassemia . the fact that iron plays a major role in the generation of ROS implies that iron chelators can also serve as antioxidants. Obviously, chelation of iron is one of the major therapeutic goals in thalassemia. Consequently, the orally administered iron chelator deferiprone was able to remove free iron from β- thalassemic red cell membranes in a dose-related fashion, Deferiprone alleviated membrane damage possibly mediated by catalytic iron, such as In a few patients with Hb E/β thalassemia in Thailand, following administration of deferiprone alone for an average of 50 weeks, Hb levels increased concomitant with a decrease in transfusion requirement One possible explanation for this finding is that deferiprone acted like an antioxidant by removing excess free iron from the cells and, as a result, ROS generation was decreased. However, the antioxidant effect of this iron chelator by itself was not sufficient to neutralize the damage induced by ROS Moreover, oral administration of other antioxidant such as vitamin E, which is a lipid antioxidant, exhibited improvement in oxidant-antioxidant balance in the plasma . Another antioxidant that acts primarily on proteins is n_acetylcysteine, which improved certain parameters resulting from oxidative damage to sickle RBCs. here we will give the N_acetylcysteine orally in dose 10mg\kg\day to the thalassemic patients for 6 months and observing its effect as antioxidant on iron overload and the frequency in blood transfusion The ultimate purpose of all these observations is to try to design a combination of antioxidants consisting of an iron chelator, such as deferiprone, vitamin E as antioxidant for the lipids, and N-acetylcysteine as antioxidant for the proteins to decrease the deleterious effect of ORS.

ELIGIBILITY:
Inclusion Criteria:

* thalassemia major children .
* On oral iron chelation .

Exclusion Criteria:

* change in the dose of iron chelation within 3 months before enrollement or during study period .
* Liver impairment
* Renal impairment
* patients not adeherent to therapy

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2024-03-23 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum ferritin level | 6 months from the baseline
  Measuring serum ferritin level (mg/dl) before and after 6 months of acetylcystein administration.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohamed YA, Meabed MH, Ashraf A, Morgan DS, Abdul Latif MG, Abd-Elkareem RM, Ahmed HM. WITHDRAWN:Randomized controlled trial of effect of N-acetylcysteine as an antioxidant on iron overload in children with thalassemia major. Clin Exp Pediatr. 2020 Nov 3. doi: 10.3345/cep.2020.00227. Online ahead of print. PMID 33147909